CLINICAL TRIAL: NCT05953974
Title: Validation of a Diagnostic Score for Encephalitis to Assess the Risk of Autoimmune Origin
Acronym: Val-Dia score
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0627
Record Dates: First submitted 2023-06-27; First posted 2023-07-20 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-06

CONDITIONS: Autoimmune Encephalitis; Autoimmune Encephalitis Caused by N-Methyl D-Aspartate Receptor Antibody (Disorder)
Keywords: Diagnostic score; auto-immune encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- NMDAr patients: Patients > or = 18 years old presenting with auto-immune encephalitis, defined according to the Graus criteria, with neuronal antibodies :
  - Anti NMDAr
  Interventions: Other: Clinical score of Granillo and al.
- LGI1 patients: Patients > or = 18 years old presenting with auto-immune encephalitis, defined according to the Graus criteria, with neuronal antibodies :
  - Anti LGI1
  Interventions: Other: Clinical score of Granillo and al.
- CASPR2 patients: Patients > or = 18 years old presenting with auto-immune encephalitis, defined according to the Graus criteria, with neuronal antibodies :
  - Anti CASPR2
  Interventions: Other: Clinical score of Granillo and al.
- GABAb patients: Patients > or = 18 years old presenting with auto-immune encephalitis, defined according to the Graus criteria, with neuronal antibodies :
  - Anti GABAb
  Interventions: Other: Clinical score of Granillo and al.
- GAD patients: Patients > or = 18 years old presenting with auto-immune encephalitis, defined according to the Graus criteria, with neuronal antibodies :
  - Anti GAD
  Interventions: Other: Clinical score of Granillo and al.

INTERVENTIONS:
Other: Clinical score of Granillo and al. — Compare the performance of the clinical prediction score of confirmed autoimmune encephalitis according to the type of antibody isolated from the CSF.

SUMMARY:
The investigators wish to test a diagnostic risk score for autoimmune encephalitis in case of encephalitis, previously validated by two American teams, in a retrospective analysis, according to the clinical and paraclinical data available in our database of the Reference Centre for Autoimmune Encephalitis and Paraneoplastic Neurological Syndromes of Professor Honnorat for patients with NMDAr, anti LGi1, anti CASPR2, anti GABAbr and anti GAD antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patient with a definite auto-immune encephalitis (Graus and al. 2016)

Exclusion Criteria:

* Uncomplete data in acute phase
* Patient with several antibodies
* Opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > or = 18 years old presenting with auto-immune encephalitis, defined according to the Graus criteria, with neuronal antibodies :
  * Anti NMDAr
  * Anti LGI1
  * Anti CASPR2
  * Anti GABAb
  * Anti GAD
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Validation of a diagnostic score for encephalitis to assess the risk of autoimmune origin. | At baseline
  Comorbidities assessed by the Charlson score
Symptoms in the acute phase | At baseline
Mode of onset of disease | At baseline
Results of lumbar puncture | At baseline
Results of antineuronal antibodies in CSF | At baseline
Results of antineuronal antibodies in serum | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France

IPD SHARING:
Plan to Share IPD: No